CLINICAL TRIAL: NCT06327425
Title: Magnetocardiography for Precise Identification of the Site of Origin of Tachyarrhythmia
Brief Title: MCG for Localization of Tachyarrhythmia's Origin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MCG-Tachyarrhythmia
Record Dates: First submitted 2024-03-11; First posted 2024-03-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-02

CONDITIONS: Tachyarrhythmia; Atrial Flutter; Paroxysmal Supraventricular Tachycardia; Atrial Tachycardia; Atrial Fibrillation; Premature Ventricular Contraction
MeSH Terms: conditions — Tachycardia; Atrial Flutter; Tachycardia, Ventricular; Atrial Fibrillation; Ventricular Premature Complexes | interventions — Magnetocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with atrial tachycardia (Experimental): Patients with atrial tachycardia will receive dynamic ECG, MCG and cardiac electrophysiologic examinations.
  Interventions: Device: Magnetocardiography
- Patients with atrial flutter (Experimental): Patients with atrial flutter will receive dynamic ECG, MCG and cardiac electrophysiologic examinations.
  Interventions: Device: Magnetocardiography

INTERVENTIONS:
Device: Magnetocardiography — Magnetocardiography

SUMMARY:
This is an exploratory research aiming to accurately identify the site of origin of tachyarrhythmia using Magnetocardiography (MCG), which will have guiding significance for early diagnosis, the formulation of treatment plans and preoperative positioning for radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-79 years old;
* Those whose conditions are comparatively stable and who have been diagnosed by an attending physician （or physicians with higher qualifications） with paroxysmal supraventricular tachycardia, atrial tachycardia, atrial flutter, atrial fibrillation, or premature ventricular contractions, and who are capable of performing MCG and cardiac electrophysiologic examinations after evaluation.
* Signed informed consent.

Exclusion Criteria:

* Those with known structural heart disease such as cardiomyopathy and valvular disease;
* Those with history of other cardiovascular diseases such as pulmonary embolism and aortic dissection;
* Those with connective tissue diseases (lupus erythematosus, rheumatoid arthritis, dermatomyositis, polyarteritis nodosa, etc.) combined with cardiac complications;
* Those with obvious abnormal thyroid function, severe anemia or other blood diseases and other diseases that obviously affect the circulating blood supply;
* Those with Obese (BMI>30kg/cm2) or underweight (BMI<18kg/cm2);
* Those with malignant tumors;
* Professional athletes, pregnant or breastfeeding women, alcoholics;
* Those with acute diseases or critical illnesses in other systems, such as acute or severe respiratory diseases, abnormal liver function or renal function, etc.;
* Those with infectious diseases or communicable diseases;
* Those who are unable or fail to perform magnetocardiography due to claustrophobia, physical impairment, etc.;
* Unable to or fail to cooperate with the corresponding research requirements.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy of MCG to detect the site of origin of Tachyarrhythmia using cardiac electrophysiology as a reference standard. | 12 month course of the disease
  Sensitivity, specificity, and area under the ROC curve are performed for assessing the efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Professor, Principal Investigator — Qliu Hospital of Shandong University
Locations (1):
- China, Shandong Qilu Hospital of Shandong University, Jinan, Shandong, China